CLINICAL TRIAL: NCT01875861
Title: Monitoring and Management for Metabolic Effects of Antipsychotics
Brief Title: Monitoring and Management for Metabolic Side Effects of Antipsychotics
Acronym: AMMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDP 08-375
Record Dates: First submitted 2013-06-05; First posted 2013-06-12 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Mental Health; Psychotic Disorders
Keywords: Antipsychotic Agents; Metabolic Syndrome; Quality Improvement
MeSH Terms: conditions — Psychological Well-Being; Psychotic Disorders; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Evidence-Based Quality Improvement plus external facilitation to promote uptake of quality improvement tools and improvement strategies available as part of a national initiative (the MIAMI Project) to disseminate recommendations, tools, and improvement strategies relevant to metabolic monitoring and management.
  Interventions: Other: Evidence-Based Quality Improvement Plus Facilitation
- Comparison (No Intervention): "Usual care," in the context of the MIAMI Project.

INTERVENTIONS:
Other: Evidence-Based Quality Improvement Plus Facilitation — The intervention involves researchers partnering with clinical stakeholders, offering tailoring in local implementation strategies to address barriers to metabolic side-effect monitoring and management. External facilitation to support, problem-solve and refine implementation will be provided for a six-month implementation phase.
  Other Names: EBQI/F
  Arms: Intervention

SUMMARY:
The purpose of this study is to test an approach for implementing guideline recommendations for assessing and managing metabolic side effects (including weight gain, diabetes, elevated lipids) in patients prescribed antipsychotic medications.

DETAILED DESCRIPTION:
Treatment of psychotic disorders consists primarily of antipsychotic medications, which are associated with metabolic side effects such as overweight/obesity, diabetes, and dyslipidemia. Expert consensus and evidence-based recommendations have been developed for assessment and management of these conditions; however, research studies show deficits and delays in metabolic monitoring for patients prescribed antipsychotics. This purpose of this study is to test a quality improvement intervention to enhance implementation of recommendations for assessing and managing metabolic side effects in patients prescribed antipsychotic medications.

Study Objectives are:

* Objective 1: To test the effect of an Evidence-Based Quality Improvement/Facilitation (EBQI/F) intervention as an augmentation to a national implementation initiative on rates of monitoring for metabolic side effects of antipsychotics in sites likely to encounter greater challenges to implementation.
* Objective 2: To test the effect of the EBQI/F intervention as an augmentation to the national implementation initiative on management of metabolic side effects of antipsychotics in sites likely to encounter greater challenges to implementation.
* Objective 3: To assess the direct costs of the EBQI/F intervention, and explore potential variations in costs of the EBQI/F intervention in sites with lower versus higher organizational challenges.

Methods This study employs a cluster randomized design with eligible study sites including VA Medical Centers with 300 patients receiving a new antipsychotic prescription in the first six months of Fiscal Year 2008. Twelve sites have been recruited and matched according to level of organizational readiness-to-change. Randomization to intervention or control group was conducted within each of the six site-pairs. Study participants include VA employees involved in the monitoring and management of patients treated with antipsychotics at participating sites. The intervention involves researchers partnering with clinical stakeholders, offering tailoring in local implementation strategies to address barriers to metabolic side-effect monitoring and management. External facilitation to support, problem-solve and refine implementation will be provided for a six-month implementation phase. The effectiveness of the EBQI/F intervention combined with the ongoing national quality improvement initiative at six sites (intervention sites) will be compared to six matched comparison sites exposed to the national quality improvement initiative alone (control sites).

ELIGIBILITY:
Inclusion Criteria:

- Providers involved in antipsychotic management or management of metabolic side effects and related conditions

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Owen, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helfrich CD, Blevins D, Smith JL, Kelly PA, Hogan TP, Hagedorn H, Dubbert PM, Sales AE. Predicting implementation from organizational readiness for change: a study protocol. Implement Sci. 2011 Jul 22;6:76. doi: 10.1186/1748-5908-6-76. PMID 21777479
- [Background] Owen RR, Drummond KL, Viverito KM, Marchant K, Pope SK, Smith JL, Landes RD. Monitoring and managing metabolic effects of antipsychotics: a cluster randomized trial of an intervention combining evidence-based quality improvement and external facilitation. Implement Sci. 2013 Oct 8;8:120. doi: 10.1186/1748-5908-8-120. PMID 24103648
- [Background] Fortney JC, Owen RR. Increasing treatment engagement for persons with serious mental illness using personal health records. Am J Psychiatry. 2014 Mar;171(3):259-61. doi: 10.1176/appi.ajp.2013.13121701. No abstract available. PMID 24585327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve sites were recruited, matched according to level of organizational readiness-to-change, and randomized to intervention/control group within each of the 6 site-pairs. Patients with a new antipsychotic medication start were identified using VA data in 6-month pre-implementation, implementation, and sustainability periods.
Pre-assignment Details: Participants were continuously entered into the study when starting a new antipsychotic treatment and were assessed up to 120 days later, thus the number of participants within each period is independent of one another and for some participants where the 120 days spanned two periods they are counted in more than one period.
Units Other Than Participants: Sites
Groups:
- Comparison: "Usual care" with access to information about QI tools and improvement strategies, but no Evidence-Based Quality Improvement or Facilitation components.
Period: Pre-implementation
Arm/Group | Intervention | Comparison
Started | 4779; 6 Sites | 3714; 6 Sites
Completed | 4779; 6 Sites | 3714; 6 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites
Period: Implementation
Arm/Group | Intervention | Comparison
Started (The number of patients within each period is independent of the number in other periods.) | 4546; 6 Sites | 3444; 6 Sites
Completed | 4546; 6 Sites | 3444; 6 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites
Period: Sustainability
Arm/Group | Intervention | Comparison
Started | 4306; 6 Sites | 3444; 6 Sites
Completed | 4306; 6 Sites | 3444; 6 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites

BASELINE CHARACTERISTICS:
Population: For each outcome measure, patients are selected when a new antipsychotic medication is prescribed. Some patients appear in more than one period (pre-implementation, implementation, sustainability); baseline characteristics are presented for the total sample (N=20,101) with rows for each period.
Units Other Than Participants: Sites
Groups:
- Intervention: Evidence-Based Quality Improvement plus external facilitation to promote uptake of QI tools and improvement strategies available as part of a national initiative (the MIAMI Project) to disseminate recommendations, QI tools, and improvement strategies relevant to metabolic monitoring and management.
  Evidence-Based Quality Improvement Plus Facilitation: The intervention involves researchers partnering with clinical stakeholders, offering tailoring in local implementation strategies to address barriers to metabolic side-effect monitoring and management. External facilitation to support, problem-solve and refine implementation will be provided for a six-month implementation phase.
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison | Total
Number analyzed (Participants) | 11335 | 8766 | 20101
Number analyzed (Sites) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The total sample size is smaller than the sum of participants in each study period because, according to the study design, patients may be selected for observation in more than one period.
  years
    Overall Sample | 54.19 (15.99) | 53.67 (16.62) | 53.93 (16.28)
    Pre-Implementation: number analyzed (Participants) | 4779 | 3714 | 8493
    Pre-Implementation | 54.51 (15.67) | 54.06 (16.18) | 54.31 (15.9)
    Implementation: number analyzed (Participants) | 4546 | 3444 | 7990
    Implementation | 53.75 (16.02) | 52.82 (16.64) | 53.35 (16.29)
    Sustainability: number analyzed (Participants) | 4306 | 3444 | 7750
    Sustainability | 53.45 (16.08) | 53.06 (16.54) | 53.28 (16.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total sample size is smaller than the sum of participants in each study period because, according to the study design, patients may be selected for observation in more than one period.
  Participants
    Overall Sample: Female | 1337 | 1027 | 2364
    Overall Sample: Male | 9998 | 7739 | 17737
    Pre-Implementation: number analyzed (Participants) | 4779 | 3714 | 8493
    Pre-Implementation: Female | 544 | 421 | 965
    Pre-Implementation: Male | 4235 | 3293 | 7528
    Implementation: number analyzed (Participants) | 4546 | 3444 | 7990
    Implementation: Female | 562 | 433 | 995
    Implementation: Male | 3984 | 3011 | 6995
    Sustainability: number analyzed (Participants) | 4306 | 3444 | 7750
    Sustainability: Female | 524 | 441 | 965
    Sustainability: Male | 3782 | 3003 | 6785
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total sample size is smaller than the sum of participants in each study period because, according to the study design, patients may be selected for observation in more than one period.
  Participants
    Overall Sample: Hispanic or Latino | 497 | 423 | 920
    Overall Sample: Not Hispanic or Latino | 10459 | 7865 | 18324
    Overall Sample: Unknown or Not Reported | 379 | 478 | 857
    Pre-Implementation: number analyzed (Participants) | 4779 | 3714 | 8493
    Pre-Implementation: Hispanic or Latino | 200 | 184 | 384
    Pre-Implementation: Not Hispanic or Latino | 4394 | 3341 | 7735
    Pre-Implementation: Unknown or Not Reported | 185 | 189 | 374
    Implementation: number analyzed (Participants) | 4546 | 3444 | 7990
    Implementation: Hispanic or Latino | 215 | 157 | 372
    Implementation: Not Hispanic or Latino | 4197 | 3101 | 7298
    Implementation: Unknown or Not Reported | 134 | 186 | 320
    Sustainability: number analyzed (Participants) | 4306 | 3444 | 7750
    Sustainability: Hispanic or Latino | 183 | 158 | 341
    Sustainability: Not Hispanic or Latino | 3986 | 3107 | 7093
    Sustainability: Unknown or Not Reported | 137 | 179 | 316
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7450 | 5828 | 13278
  Black | 2791 | 2239 | 5030
  Other | 398 | 206 | 604
  Unknown | 696 | 493 | 1189
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11335 | 8766 | 20101

OUTCOME MEASURES:

1. Primary Outcome: Change in Site-level Rates of Weight Monitoring at Baseline (Within 30 Days of a New Antipsychotic Prescription)
Description: For each monthly observation: The proportion of patients at each site due for weight monitoring at baseline who have weight recorded in the electronic health record.
Time Frame: Change in monitoring rates will be measured monthly through 6-month pre-implementation, implementation, and sustainability phases
Population: All patients who met inclusion criteria for this measure. Note that total for Outcome 1 is less than overall total N because patients were included for each measure independently if they met criteria any time in the 6-month implementation phases. Slightly more patients met criteria for the "follow-up monitoring" measures than "baseline monitoring."
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 9214 | 7213
Participants
  Pre-Implementation: number analyzed (Participants) | 3200 | 2516
  Pre-Implementation | 1811 | 1410
  Implementation: number analyzed (Participants) | 3118 | 2379
  Implementation | 1598 | 1109
  Sustainability: number analyzed (Participants) | 2896 | 2318
  Sustainability | 1384 | 1043
Statistical Analysis 1: Comparison: Intervention vs Comparison; Because of data discontinuity, assumptions for time series analysis did not hold. Repeated measures regression models were developed to compare overall weight monitoring rates at baseline across the implementation phases; Test type: Superiority; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.02 to 1.38]

2. Secondary Outcome: Change in Site-level Rates of Weight Monitoring at Follow-up (From 31-120 Days After a New Antipsychotic Prescription)
Description: For each monthly observation: The proportion of patients at each site due for weight monitoring at follow-up who have weight recorded in the electronic health record.
Time Frame: as for outcome 1
Population: All patients meeting inclusion/exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 9302 | 7174
Participants
  Pre-Implementation: number analyzed (Participants) | 3264 | 2532
  Pre-Implementation | 1696 | 1337
  Implementation: number analyzed (Participants) | 3141 | 2315
  Implementation | 1477 | 1005
  Sustainability: number analyzed (Participants) | 2897 | 2327
  Sustainability | 1265 | 992
Statistical Analysis 1: Comparison: Intervention vs Comparison; See comments about time series analysis for primary outcome measure. Repeated measures regression analysis of the likelihood of monitoring for each time period was conducted; Test type: Superiority; Odds Ratio (OR) = 1.2, 95% CI 2-sided [1.03 to 1.39]

3. Secondary Outcome: Change in Site-level Rates of Management for Obesity or Weight Gain Within 30 Days After a Recording of 5% Gain in Body Weight
Description: For each monthly observation: The proportion of patients at each site with weight gain that have guideline-recommended weight management (e.g., counseling about diet or exercise, referral to weight management program) initiated within 30 days.
Time Frame: Change in weight management rates will be measured monthly through 6-month pre-implementation, implementation, and sustainability phases
Population: All patients meeting inclusion/exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 586 | 379
Participants
  Pre-Implementation: number analyzed (Participants) | 149 | 108
  Pre-Implementation | 25 | 23
  Implementation: number analyzed (Participants) | 232 | 116
  Implementation | 46 | 28
  Sustainability: number analyzed (Participants) | 205 | 155
  Sustainability | 50 | 65

ADVERSE EVENTS:
Arm/Group | Intervention | Comparison
Serious Adverse Events (participants affected / at risk) | 0/11335 | 0/8766
Other Adverse Events (participants affected / at risk) | 0/11335 | 0/8766

LIMITATIONS AND CAVEATS:
This study was planned in conjunction with a national effort to improve metabolic monitoring and management for Veterans prescribed antipsychotic medications. However, this study's implementation activities started after the national effort ended..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes